CLINICAL TRIAL: NCT06066684
Title: Prediction Modelling of TKA Non-responders Using Clinical and Pain Sensitization Measures
Brief Title: Pain Phenotyping in Knee OA: a Pilot Trial
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: CTO3624
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-09

CONDITIONS: Osteo Arthritis Knee; Chronic Post-operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: n/a, observational — n/a, observational study

SUMMARY:
Osteoarthritis (OA) is disease in which the joint breaks down, causing pain. The decision to surgically replace the knee, a procedure called total knee arthroplasty (TKA), depends on x-ray results as well as pain and dysfunction. Despite TKA resulting in good outcomes for most patients, between 1 in 10 and 1 in 5 patients remain in significant pain - i.e., are 'TKA non-responders'. Two pain conditions - myofascial pain syndrome (MPS) and central sensitization - frequently coexist with signs of OA and may contribute to a TKA non-responder profile. MPS, caused by knots within skeletal muscle, can contribute to an OA patient's pain and dysfunction. In central sensitization, faulty pain sensing leads to increased pain sensitivity. However, there is currently no established process to identify these sources of pain and potential associated TKA non-responder risk. Our research aims conduct a pilot study to examine the impact of pain diagnosis tools to help orthopedic surgeons identify potential TKA nonresponders. This new approach may increase healthcare efficiency (reduce TKA waitlist and length of hospital stay), and help patients receive the right care at the right time.

ELIGIBILITY:
Inclusion Criteria:

* adult patients aged 18 or older
* on the waitlist for TKA (unilateral) for knee osteoarthritis

Exclusion Criteria:

* undergoing revision or non-elective surgery
* unable to provide informed consent and follow study procedures

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: adult knee osteoarthritis patients
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2025-06-18 (Estimated); Study Completion 2025-09-18 (Estimated)

PRIMARY OUTCOMES:
Clinical prediction model feasibility as determined by: Recruitment rate, follow-up at 12 months post-op, multivariable logistic regression | 21 months

SECONDARY OUTCOMES:
Pain regions and pain pattern, as assessed by Pain Body Diagram | 21 months
Likelihood of neuropathic pain component, as assessed by the painDETECT questionnaire | 21 months
Symptoms of central sensitisation, as assessed by the Central Sensitization Inventory questionnaire | 21 months
Physical function, as assessed by the Aggregate Locomotor Function test | 21 months
Prevalence of myofascial trigger points | 21 months
Pain facilitation, as assessed by Temporal Summation of Pain (wind-up) | 21 months
Deep tissue pain sensitivity, as assessed by Pain Pressure Threshold | 21 months

CONTACTS AND LOCATIONS:
Overall Officials: Dinesh Kumbhare, MD, PhD, Principal Investigator — UHN
Locations (2):
- Canada (2):
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Toronto Western Hospital, Toronto, Ontario